CLINICAL TRIAL: NCT00736125
Title: A Comparison of Intraoperative Embolic Events During Total Knee Arthroplasty Performed With CarboJet Assisted Versus Standard Orthopedic Techniques: A Pilot Study
Brief Title: A Study to Determine if Carbon Dioxide Lavage During Total Knee Surgery Reduces Intraoperative Embolic Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kinamed Incorporated (Industry)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01226
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Results first posted 2013-04-18 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Complications; Memory Disorders
Keywords: postoperative cognitive dysfunction; total knee arthroplasty; cerebral emboli; carbon dioxide lavage; pulsatile saline lavage
MeSH Terms: conditions — Postoperative Complications; Memory Disorders; Postoperative Cognitive Complications; Intracranial Embolism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Device: pulsatile saline lavage
- 2 (Active Comparator)
  Interventions: Device: carbon dioxide lavage

INTERVENTIONS:
Device: pulsatile saline lavage — Prior to cement application, cut bone surfaces are cleaned using pulsatile saline lavage
  Arms: 1
Device: carbon dioxide lavage — Prior to cement application, cut bone surfaces are cleaned using carbon dioxide lavage
  Arms: 2

SUMMARY:
The purpose of this study is to determine if the use of a carbon dioxide lavage device (CarboJet) to clean bone surfaces during total knee surgery decreases intraoperative embolic events when compared with standard orthopedic techniques.

DETAILED DESCRIPTION:
Elderly patients undergoing major, orthopedic surgery are at risk of developing postoperative cognitive dysfunction (POCD) or memory impairment following surgery. Transcranial doppler (TCD) monitoring of blood flow to the brain has detected cerebral emboli in 60% of patients following release of the thigh tourniquet during total knee replacement or arthroplasty (TKA). These cerebral embolic events may represent one of the mechanisms responsible for postoperative cognitive problems.

The standard surgical technique for TKA involves cleaning the bone surfaces with pulsed saline lavage prior to cementation and prosthesis insertion. The CarboJet Assisted technique utilizes carbon dioxide lavage to clean and dry the femur canal and bone surfaces prior to cementation and implantation. Because it removes fat globules and marrow particulates from the bone surfaces, it is hypothesized that the use of a carbon dioxide lavage technique in TKA will result in fewer thromboembolic events and increased cement penetration compared with the standard technique using pulsed saline lavage. Cement penetration affects the strength of the bone-cement interface and, therefore, contributes to implant longevity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 50 years or older who are scheduled for elective TKA with a cemented Smith and Nephew Prosthesis design

Exclusion Criteria:

* Dementia or severe cognitive impairment
* Severe visual or hearing impairments
* Inability to follow directions or comprehend the English language
* Females who are pregnant
* Abnormal distal femur geometry
* Pre-existing hardware or abnormal bony architecture in the proximal tibia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terri G Monk, MD, Principal Investigator — Duke University
Locations (1):
- Veterans Affairs Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: during pre-op workup for TKA, patients were informed about study and asked if they wanted to participate.
Groups:
- 1 Pulsatile Saline Lavage: pulsatile saline lavage : Prior to cement application, cut bone surfaces are cleaned using pulsatile saline lavage
- 2 Carbon Dioxide Lavage: carbon dioxide lavage : Prior to cement application, cut bone surfaces are cleaned using carbon dioxide lavage
Period: Overall Study
Arm/Group | 1 Pulsatile Saline Lavage | 2 Carbon Dioxide Lavage
Started | 10 | 10
Completed | 9 | 8
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Pulsatile Saline Lavage | 2 Carbon Dioxide Lavage | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (3.3) | 63.9 (3.7) | 63.1 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Number of Cerebral Emboli During Surgery as Measured by Transcranial Doppler (TCD)
Time Frame: During surgery
Measure: Number; unit: emboli
Arm/Group | 1 Pulsatile Saline Lavage | 2 Carbon Dioxide Lavage
Number analyzed (Participants) | 7 | 6
emboli | 0 | 3

2. Secondary Outcome: Number of Patients With Emboli in the High Category
Time Frame: During surgery
Measure: Number; unit: Patients w/ emboli in high category
Arm/Group | 1 Pulsatile Saline Lavage | 2 Carbon Dioxide Lavage
Number analyzed (Participants) | 9 | 8
Patients w/ emboli in high category | 9 | 5

3. Secondary Outcome: Number of Patients With Delirium During Hospital Stay
Time Frame: First 3 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | 1 Pulsatile Saline Lavage | 2 Carbon Dioxide Lavage
Number analyzed (Participants) | 10 | 10
Participants | 1 | 4
Statistical Analysis 1: Comparison: 1 Pulsatile Saline Lavage vs 2 Carbon Dioxide Lavage; Test type: Equivalence — nonparametric data were analyzed using Mann Whitney U Tests; p > 0.05, t-test, 2 sided

4. Other Pre Specified Outcome: Changes in Neurocognitive Tests Following Surgery
Description: Hopkins Verbal Learning Test (HVLT).This is a test of verbal learning and memory.
  The scale is the number of words retained. The total score for the test administered ranges from 0 to 12. Higher values represent better outcomes.
Time Frame: 3 months following surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 1 Pulsatile Saline Lavage | 2 Carbon Dioxide Lavage
Number analyzed (Participants) | 9 | 10
score on a scale | 1.67 (1.6) | 4.7 (1.5)
Statistical Analysis 1: Comparison: 1 Pulsatile Saline Lavage vs 2 Carbon Dioxide Lavage; Test type: Superiority; p > 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | 1 Pulsatile Saline Lavage | 2 Carbon Dioxide Lavage
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No